CLINICAL TRIAL: NCT06224621
Title: Percutaneous Endocardial Septal Radiofrequency Ablation in the Treatment of Obstructive Hypertrophic Cardiomyopathy: a Prospective, Multicenter, Single-arm Objective Performance Criteria Trial
Brief Title: Percutaneous Endocardial Septal Radiofrequency Ablation in Obstructive Hypertrophic Cardiomyopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-ZX012
Record Dates: First submitted 2024-01-02; First posted 2024-01-25 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-01

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Percutaneous Endocardial Septal Radiofrequency Ablation (PESA) is used to ablatethe hypertrophied septum of obstructive hypertrophic cardiomyopathy (oHCM) patients.
  Interventions: Procedure: Percutaneous Endocardial Septal Radiofrequency Ablation

INTERVENTIONS:
Procedure: Percutaneous Endocardial Septal Radiofrequency Ablation — Percutaneous Endocardial Septal Radiofrequency Ablation (PESA) is used to ablatethe hypertrophied septum of obstructive hypertrophic cardiomyopathy (oHCM) patients.

SUMMARY:
This prospective, multicenter, single-arm objective performance criteria trial is designed to assess the efficacy and safety of the Percutaneous Endocardial Septal Radiofrequency Ablation (PESA) procedure in the treatment of obstructive hypertrophic cardiomyopathy (oHCM). The primary objectives include investigating:

1. the treatment efficacy and safety of PESA treatment in oHCM patients with either left ventricular outflow tract obstruction (LVOTO) or midventricular obstruction;
2. the impact of PESA treatment on the functional capacity, quality of life and long-term prognosis of oHCM patients with either LVOTO or midventricular obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of hypertrophic cardiomyopathy;
* At least 18 years old;
* The presence of a resting or maximum provoked LVOT/midventricular gradient of ≥50 mmHg with symptoms, despite maximum tolerated medical therapy;
* Willing to receive PESA treatment;
* LVEF≥55%;
* Signed and dated written informed consent and willing to return for clinical follow-up.

Exclusion Criteria:

* Midventricular obstruction rendered by isolated papillary muscle hypertrophy;
* Complete right bundle branch block;
* Acute decompensation heart failure with NYHA IV;
* Previous septal reduction therapy including surgical and interventional procedures;
* Combination of other diseases requiring surgical treatment (including but not limited to coronary artery bypass grafting and apical aneurysm);
* Contraindications of radiofrequency ablation procedure;
* Women who are pregnant or lactating, or who plan to become pregnant while in the trial;
* Currently enrolled in another investigational device or drug trial;
* Combining any other clinical condition with a life expectancy less than 1 year.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in LVOT gradiant/midventricular gradient | 6 months,9 months and 12 months
  Change in Left ventricular outflow tract gradient pre- and post- intervention

SECONDARY OUTCOMES:
Change in 6 minute walking test | 6 months,9 months and 12 months
  Change in 6 minute walking distance pre- and post- intervention
Change in NYHA cardiac function class | 6 months,9 months and 12 months
  A system used to categorize the severity of heart failure based on the functional limitations of individuals.
Change in cTnT | 6 months,9 months and 12 months
  Cardiac biomarker
Change in cTnI | 6 months,9 months and 12 months
  Cardiac biomarker
Change in NT-proBNP | 6 months,9 months and 12 months
  Cardiac biomarker
Change in Participant-reported Health-related Quality of Life as Assessed by the KCCQ Score | 6 months,9 months and 12 months
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a patient reported outcome instrument with minimum score = 0 and maximum score = 100 where higher score indicates better health status. There are no units to the score. The instrument utilizes a recall period of 2 weeks over which patients describe the frequency and severity of their symptoms, their physical and social limitations, and how they perceive their heart failure symptoms to affect their quality of life. quality of life
Change in Left ventricular ejection fraction (LVEF) | 6 months,9 months and 12 months
  LVEF measured by echocardiography
Change in Left ventricular end-diastolic diameter (LVEDD) | 6 months,9 months and 12 months
  LVEDD measured by echocardiography
Change in Left atrial diameter (LAD) | 6 months,9 months and 12 months
  LAD measured by echocardiography
Change in Maximal wall thickness (MWT) | 6 months,9 months and 12 months
  MWT measured by echocardiography
Change in Left ventricular mass index (LVMi) | 6 months,9 months and 12 months
  LVMi measured by cardiac magnetic resonance
Change in Late gadolinium enhancement (LGE) | 6 months,9 months and 12 months
  LGE measured by cardiac magnetic resonance
Change in Cardiac index (CI) | 6 months,9 months and 12 months
  CI measured by cardiac magnetic resonance

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, National Centre for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF